CLINICAL TRIAL: NCT05143671
Title: Prospective Evaluation for Hybrid Cardiac Procedures
Acronym: PERHAPS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Bruno, Clinical Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3959
Record Dates: First submitted 2021-11-05; First posted 2021-12-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Left Main Coronary Artery Disease; Left Anterior Descending Coronary Artery Stenosis; Valve Disease, Heart; Carotid Stenosis; Coronary Artery Disease; Heart Diseases; Heart Valve Diseases; Carotid Occlusion
Keywords: coronary artery disease; carotid stenosis; percutaneous coronary intervention; coronary artery bypass; carotid artery diseases; heart valves; stent
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Carotid Stenosis; Heart Diseases; Carotid Artery Diseases | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Hybrid coronary revascularization strategy (HCR): Patients who undergo a combination of coronary artery bypass grafting and PCI.
  Interventions: Procedure: Coronary artery bypass grafting; Procedure: Percutaneous coronary intervention
- Hybrid valve and coronary disease correction: Patients who undergo a combination of surgical valve replacement and PCI.
  Interventions: Procedure: Percutaneous coronary intervention; Procedure: Surgical valve replacement
- Hybrid coronary and carotid artery disease treatment: Patients who undergo a combination of coronary artery bypass grafting and carotid stenting.
  Interventions: Procedure: Coronary artery bypass grafting; Procedure: Carotid artery stenting

INTERVENTIONS:
Procedure: Coronary artery bypass grafting — Coronary artery bypass grafting in coronary revascularization.
  Groups: Hybrid coronary and carotid artery disease treatment; Hybrid coronary revascularization strategy (HCR)
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention in coronary revascularization.
  Groups: Hybrid coronary revascularization strategy (HCR); Hybrid valve and coronary disease correction
Procedure: Surgical valve replacement — Surgical mitral and / or aortic valve replacement.
  Groups: Hybrid valve and coronary disease correction
Procedure: Carotid artery stenting — Carotid artery stenting.
  Groups: Hybrid coronary and carotid artery disease treatment

SUMMARY:
Multidisciplinary team-approach in order to offer personalized treatments represents the emerging mainstream in cardiovascular medicine. "Hybrid operative rooms" allow to offer selected heart-disease patients truly "tailored" operations.

This study wants to evaluate the effectiveness and safety of Hybrid Procedures in cardiac patients in three subgroups of patients:

* Hybrid coronary revascularization strategy (coronary by-pass + PCI);
* Hybrid valve and coronary disease correction (combination of surgical valve replacement and PCI);
* Hybrid coronary and carotid artery disease treatment (combination of coronary by-pass and carotid stenting).

The investigators hypothesize that morbidity might be reduced by 50% in hybrid procedures group as compared with predicted Society of Thoracic Surgery (STS) score.

DETAILED DESCRIPTION:
Cardiovascular medicine is actually evolving fast and multidisciplinary team-approach in order to offer personalized treatments represents the emerging mainstream. The possibility to realize combinations of treatments traditionally available only in the catheterization laboratory and in the operating room represent the rationale for "hybrid operative rooms" facilities allowing to offer selected heart-disease patients truly "tailored" operations. Such "Hybrid" management strategies usually combine transcatheter techniques and surgery (often minimally invasive) in order to combine the reduced invasiveness of the former with the effectiveness of the latter. Common examples of surgical and transcatheter combinations are: hybrid revascularization performed with coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI); combined heart valve and coronary disease treated with valve surgery and PCI; combined endo- and epicardial ablation of atrial fibrillation; thoracic aneurysms treated with endovascular stenting and surgical debranching of the arch; carotid artery stenting along with CABG. Given the relatively recent development of these techniques, indications and patient selection are yet to be defined and a productive collaboration between surgeons and interventional cardiologists is of paramount importance.

Aim of the study is to evaluate the effectiveness and safety of Hybrid Procedures in cardiac patients. Specifically, three subgroups will be analysed:

* Hybrid coronary revascularization strategy (HCR, coronary by-pass + PCI);
* Hybrid valve and coronary disease correction (combination of surgical valve replacement and PCI);
* Hybrid coronary and carotid artery disease treatment (combination of coronary by-pass and carotid stenting).

The local Heart Team (cardiac surgeon, interventional cardiologist, clinical cardiologist and anaesthetist) will decide which patients will be referred for hybrid treatment. Typically, this happens when the Heart Team feels that hybrid treatment could reduce the overall risk of a combined procedure.

The patient population consists of adult patients with:

* Multi-vessel coronary artery disease (CAD) involving the left main and/or the left anterior descending artery with indication for revascularization;
* Severe, symptomatic valvular disease and CAD with indication for revascularization;
* Significant unilateral carotid stenosis and CAD with indication for revascularization.

In a previous data review board on the Heart Team activity, we recognized that 10% of discussed patients are referred for hybrid procedures (HP) and that observed operative mortality was strongly lower than that predicted by STS and EuroSCORE (2.5% versus 10.1% and 5.9%, respectively). Morbidity was not prospectively investigated. For sample size estimation, the investigators hypothesized that Morbidity might be reduced by 50% in HP group as compared with predicted STS. The mean expected STS morbidity estimated in the study population is 32.57%. Accordingly, a total number of 111 patients with an alpha error of 5% and a beta error of 20% has been calculated to be needed to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, inclusive of release of medical information
* Age ≥ 18 years
* CAD with indication for revascularization
* Coronary anatomy as follows:

  * Multivessel-CAD involving the left anterior descending (LAD) (proximal or mid) and/or the left main (LM) (ostial, mid-shaft or distal) with at least one further epicardial coronary artery requiring treatment (LCX or RCA), OR
  * Single vessel disease involving the LAD and a major diagonal, both requiring independent revascularization with at least one stent
* Severe aortic stenosis/insufficiency and/or mitral stenosis/insufficiency requiring surgery, with CAD (involving one or more vessels), suitable for PCI
* CAD with indication for revascularization with severe unilateral carotid stenosis (>85%)
* Ability to tolerate, and no plans to interrupt dual antiplatelet therapy (DAPT) for:

  * At least 6 months in presentation was stable CAD,
  * At least 12 months if presentation was a biomarker-positive acute coronary syndrome (ACS)
* Willing to comply with the follow-up required by the protocol.

Exclusion Criteria:

* Previous cardiac surgery of any kind
* Previous thoracic surgery involving the left pleural space (if a left thoracotomy approach is planned)
* Complicated or unsuccessful PCI within 30 days prior
* Total occlusion (TIMI 0 or 1 flow) of the LM or LAD
* Cardiogenic shock at time of screening
* Any prior lung resection
* End-stage renal disease on dialysis
* Extra-cardiac illness that is expected to limit survival to less then 5 years
* Allergy or hypersensitivity to any of the study drugs or devices used in protocol
* Patient unable to give informed consent or potentially noncompliant with the study protocol, in the judgement of the investigator
* Pregnant at time of screening, or unwilling to use effective birth control measures while dual antiplatelet therapy is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with:
  * Multi-vessel CAD involving the laft main (LM) and/or the left anterior descending (LAD) artery with indication for revascularization;
  * Severe, symptomatic valvular disease and CAD with indication for revascularization;
  * Significant unilateral carotid stenosis and CAD with indication for revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with stroke | 6 days after operation
  Rapid onset of a new neurological deficit attributed to an obstruction in cerebral blood flow and/or cerebral hemorrhage with no apparent non-vascular cause (e.g., trauma, tumor, or infection) that i) persists beyond 24 hours, or ii) less than 24 hours if: a) associated with infarction or hemorrhage on an imaging study, or b) treated with pharmacologic or mechanical intervention, or c) results in death.
Number of participants with renal failure | 6 days after operation
  Acute or worsening renal failure resulting in one or more of the following: 1. Increase of serum creatinine to ≥ 4.0 with an increase of at least 0.5mg/dl or 3x most recent preoperative creatinine level. 2. A new requirement for dialysis postoperatively.
Number of participants with prolonged ventilation > 24 hours | 25 hours after operative room exit.
  Prolonged postoperative pulmonary ventilation > 24.0 hours.
Number of participants with deep sternal wound infection | Diagnosis within 30 days of the operation or >30 days after procedure but during hospital stay for surgery.
  Deep sternal wound infection or mediastinitis (according to Centers for Disease Control (CDC) definition)
Number of participants who undergo reoperation | 6 days after operation
  Reoperation for bleeding/tamponade, valvular dysfunction, graft failure, aortic reintervention, or other cardiac reason.
Number of participants with major morbidity or operative mortality | 6 days after operation
  A composite endpoint defined as any of the outcomes listed in the first six rows of this list
Number of participants with short stay | 6 days after operation
  Patient length of stay < 6 days. Discharged alive and within 5 days of surgery
Number of participants with long stay | 15 days after operation
  Patient length of stay > 14 days. Failure to be discharged within 14 days of surgery

SECONDARY OUTCOMES:
Cardiovascular events | 30 days post procedure and 12 months
  Cardiovascular events include: individual components of major adverse cardiac and cerebrovascular events (MACCE) (all-cause mortality, ischemic stroke, miocardial infarction, unplanned revascularization), ischemia-driven revascularization, cardiovascular and non-cardiovascular mortality, stent thrombosis, symptomatic graft stenosis or occlusion, re-hospitalization and othe medical encounters (all-cause and cardiovascular).
Bleeding | 30 days post procedure and 12 months
  Site assessed bleeding complications will be reported using the Bleeding Academic Research Consortium Scale. This scale ranges from Type 0 bleeding to Type 5 b bleeding. The higher the score is, the worse the outcome is.
Rate of one or more additional adverse event. | 30 days post procedure and 12 months
  Rate of one or more additional adverse event among this list:
  * Acute renal failure or worsening renal function resulting in one or both of the following: increase in serum creatinine by ≥0.5 mg/dL or ≥25% from baseline, or need for dialysis.
  * Atrial fibrillation requiring treatment (including drug therapy, cardioversion or ablation procedures).
  * Major arrhythmia (any supraventricular tachycardia requiring cardioversion, ventricular tachycardia or fibrillation requiring treatment, or bradyarrhythmia requiring temporary or permanent pacemaker).
  * Sternal wound dehiscence.
  * Infection requiring intravenous antibiotics for treatment.
  * Intubation lenght >48 hours.
  * Respiratory failure defined as continued mechanical ventilation required for greater than 48 hours post operatively.
  * Post-pericardiotomy syndrome: an inflammatory response to cardiothoracic surgery.
Health Status through angina assessment. | 30 days post procedure and 12 months
  Angina class measured by the Canadian Cardiovascular Society class. This class ranges from class I to class IV. The higher the class is, the worse the outcome is.
Health Status through quality of life assessment. | 30 days post procedure and 12 months
  Quality of Life will be measured, using the Short Form-12 (SF-12) general health status questionnaire and EuroQoL 5-D (EuroQoL) questionnaire, which measures health state preference from the individual and societal perspective.
Cost-effectiveness | 12 months post procedure
  Overall costs of hospitalization and quality-adjusted life expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Piergiorgio Bruno, MD, Principal Investigator
Locations (1):
- IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Byrne JG, Leacche M, Vaughan DE, Zhao DX. Hybrid cardiovascular procedures. JACC Cardiovasc Interv. 2008 Oct;1(5):459-68. doi: 10.1016/j.jcin.2008.07.002. PMID 19463346
- [Background] Leacche M, Umakanthan R, Zhao DX, Byrne JG. Surgical update: hybrid procedures, do they have a role? Circ Cardiovasc Interv. 2010 Oct;3(5):511-8. doi: 10.1161/CIRCINTERVENTIONS.110.957951. No abstract available. PMID 20959598
- [Background] Loop FD, Lytle BW, Cosgrove DM, Stewart RW, Goormastic M, Williams GW, Golding LA, Gill CC, Taylor PC, Sheldon WC, et al. Influence of the internal-mammary-artery graft on 10-year survival and other cardiac events. N Engl J Med. 1986 Jan 2;314(1):1-6. doi: 10.1056/NEJM198601023140101. PMID 3484393
- [Background] Diegeler A, Thiele H, Falk V, Hambrecht R, Spyrantis N, Sick P, Diederich KW, Mohr FW, Schuler G. Comparison of stenting with minimally invasive bypass surgery for stenosis of the left anterior descending coronary artery. N Engl J Med. 2002 Aug 22;347(8):561-6. doi: 10.1056/NEJMoa013563. PMID 12192015
- [Background] Lytle BW, Cosgrove DM, Loop FD, Borsh J, Goormastic M, Taylor PC. Perioperative risk of bilateral internal mammary artery grafting: analysis of 500 cases from 1971 to 1984. Circulation. 1986 Nov;74(5 Pt 2):III37-41. PMID 3490331
- [Background] Tatoulis J, Buxton BF, Fuller JA. Patencies of 2127 arterial to coronary conduits over 15 years. Ann Thorac Surg. 2004 Jan;77(1):93-101. doi: 10.1016/s0003-4975(03)01331-6. PMID 14726042
- [Background] Ben-Gal Y, Mohr R, Braunstein R, Finkelstein A, Hansson N, Hendler A, Moshkovitz Y, Uretzky G. Revascularization of left anterior descending artery with drug-eluting stents: comparison with minimally invasive direct coronary artery bypass surgery. Ann Thorac Surg. 2006 Dec;82(6):2067-71. doi: 10.1016/j.athoracsur.2006.06.041. PMID 17126111
- [Background] Fraund S, Herrmann G, Witzke A, Hedderich J, Lutter G, Brandt M, Boning A, Cremer J. Midterm follow-up after minimally invasive direct coronary artery bypass grafting versus percutaneous coronary intervention techniques. Ann Thorac Surg. 2005 Apr;79(4):1225-31. doi: 10.1016/j.athoracsur.2004.08.082. PMID 15797053
- [Background] Alexander JH, Hafley G, Harrington RA, Peterson ED, Ferguson TB Jr, Lorenz TJ, Goyal A, Gibson M, Mack MJ, Gennevois D, Califf RM, Kouchoukos NT; PREVENT IV Investigators. Efficacy and safety of edifoligide, an E2F transcription factor decoy, for prevention of vein graft failure following coronary artery bypass graft surgery: PREVENT IV: a randomized controlled trial. JAMA. 2005 Nov 16;294(19):2446-54. doi: 10.1001/jama.294.19.2446. PMID 16287955
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Harskamp RE, Zheng Z, Alexander JH, Williams JB, Xian Y, Halkos ME, Brennan JM, de Winter RJ, Smith PK, Lopes RD. Status quo of hybrid coronary revascularization for multi-vessel coronary artery disease. Ann Thorac Surg. 2013 Dec;96(6):2268-77. doi: 10.1016/j.athoracsur.2013.07.093. PMID 24446561
- [Background] Mauri L, Orav EJ, Kuntz RE. Late loss in lumen diameter and binary restenosis for drug-eluting stent comparison. Circulation. 2005 Jun 28;111(25):3435-42. doi: 10.1161/CIRCULATIONAHA.104.513952. Epub 2005 Jun 20. PMID 15967844
- [Background] Leacche M, Byrne JG, Solenkova NS, Reagan B, Mohamed TI, Fredi JL, Zhao DX. Comparison of 30-day outcomes of coronary artery bypass grafting surgery verus hybrid coronary revascularization stratified by SYNTAX and euroSCORE. J Thorac Cardiovasc Surg. 2013 Apr;145(4):1004-1012. doi: 10.1016/j.jtcvs.2012.03.062. Epub 2012 Apr 25. PMID 22541514
- [Background] Harskamp RE, Brennan JM, Xian Y, Halkos ME, Puskas JD, Thourani VH, Gammie JS, Taylor BS, de Winter RJ, Kim S, O'Brien S, Peterson ED, Gaca JG. Practice patterns and clinical outcomes after hybrid coronary revascularization in the United States: an analysis from the society of thoracic surgeons adult cardiac database. Circulation. 2014 Sep 9;130(11):872-9. doi: 10.1161/CIRCULATIONAHA.114.009479. Epub 2014 Jul 23. PMID 25055814
- [Background] Verhaegh AJ, Accord RE, van Garsse L, Maessen JG. Hybrid coronary revascularization as a safe, feasible, and viable alternative to conventional coronary artery bypass grafting: what is the current evidence? Minim Invasive Surg. 2013;2013:142616. doi: 10.1155/2013/142616. Epub 2013 Apr 3. PMID 23691303
- [Background] Wrigley BJ, Dubey G, Spyt T, Gershlick AH. Hybrid revascularisation in multivessel coronary artery disease: could a combination of CABG and PCI be the best option in selected patients? EuroIntervention. 2013 Mar;8(11):1335-41. doi: 10.4244/EIJV8I11A202. No abstract available. PMID 23538160
- [Background] Green KD, Lynch DR Jr, Chen TP, Zhao D. Combining PCI and CABG: the role of hybrid revascularization. Curr Cardiol Rep. 2013 Apr;15(4):351. doi: 10.1007/s11886-013-0351-9. PMID 23420447
- [Background] Santana O, Funk M, Zamora C, Escolar E, Lamas GA, Lamelas J. Staged percutaneous coronary intervention and minimally invasive valve surgery: results of a hybrid approach to concomitant coronary and valvular disease. J Thorac Cardiovasc Surg. 2012 Sep;144(3):634-9. doi: 10.1016/j.jtcvs.2011.11.008. Epub 2011 Dec 10. PMID 22154788
- [Background] Santana O, Pineda AM, Cortes-Bergoderi M, Mihos CG, Beohar N, Lamas GA, Lamelas J. Hybrid approach of percutaneous coronary intervention followed by minimally invasive valve operations. Ann Thorac Surg. 2014 Jun;97(6):2049-55. doi: 10.1016/j.athoracsur.2014.02.039. Epub 2014 Apr 13. PMID 24725838
- [Background] Byrne JG, Leacche M, Unic D, Rawn JD, Simon DI, Rogers CD, Cohn LH. Staged initial percutaneous coronary intervention followed by valve surgery ("hybrid approach") for patients with complex coronary and valve disease. J Am Coll Cardiol. 2005 Jan 4;45(1):14-8. doi: 10.1016/j.jacc.2004.09.050. PMID 15629366
- [Background] Versaci F, Reimers B, Del Giudice C, Schofer J, Giacomin A, Sacca S, Gandini R, Albiero R, Pellegrino A, Bertoldo F, Simonetti G, Chiariello L. Simultaneous hybrid revascularization by carotid stenting and coronary artery bypass grafting: the SHARP study. JACC Cardiovasc Interv. 2009 May;2(5):393-401. doi: 10.1016/j.jcin.2009.02.010. PMID 19463460
- [Background] Velissaris I, Kiskinis D, Anastasiadis K. Synchronous carotid artery stenting and open heart surgery. J Vasc Surg. 2011 May;53(5):1237-41. doi: 10.1016/j.jvs.2010.11.049. Epub 2011 Jan 17. PMID 21247729
- [Background] Chiariello L, Nardi P, Pellegrino A, Saitto G, Chiariello GA, Russo M, Zeitani J, Versaci F. Simultaneous carotid artery stenting and heart surgery: expanded experience of hybrid surgical procedures. Ann Thorac Surg. 2015 Apr;99(4):1291-7. doi: 10.1016/j.athoracsur.2014.11.043. Epub 2015 Feb 7. PMID 25661578
- [Background] Mendiz OA, Fava CM, Lev GA, Valdivieso LR, Caponi G, Hidalgo Alava GF, Favaloro RR. Hybrid strategy for unstable patients with severe carotid and cardiac disease requiring surgery. Cardiol J. 2015;22(1):25-30. doi: 10.5603/CJ.a2014.0001. Epub 2014 Feb 14. PMID 24526504
- [Background] Chiariello L, Tomai F, Zeitani J, Versaci F. Simultaneous hybrid revascularization by carotid stenting and coronary artery bypass grafting. Ann Thorac Surg. 2006 May;81(5):1883-5. doi: 10.1016/j.athoracsur.2005.04.086. PMID 16631695
- [Background] Wu H, Sun H, Jiang X, Ma W, Wang X, Zhang J, Hu S. Simultaneous hybrid revascularization by peripheral artery stenting and off-pump coronary artery bypass: the early results. Ann Thorac Surg. 2011 Mar;91(3):661-4. doi: 10.1016/j.athoracsur.2010.10.057. PMID 21352975
- [Background] Yang T, Zhang L, Wang X, Dong H, Jiang X, Sun H. Revascularization by carotid artery stenting and off-pump coronary artery bypass. ANZ J Surg. 2016 Jul;86(7-8):602-7. doi: 10.1111/ans.12586. Epub 2014 Apr 3. PMID 24698016
- [Background] Van der Heyden J, Van Neerven D, Sonker U, Bal ET, Kelder JC, Plokker HW, Suttorp MJ. Carotid artery stenting and cardiac surgery in symptomatic patients. JACC Cardiovasc Interv. 2011 Nov;4(11):1190-6. doi: 10.1016/j.jcin.2011.07.012. PMID 22115658
- [Background] Versaci F, Del Giudice C, Scafuri A, Zeitani J, Gandini R, Nardi P, Salvati A, Pampana E, Sebastiano F, Romagnoli A, Simonetti G, Chiariello L. Sequential hybrid carotid and coronary artery revascularization: immediate and mid-term results. Ann Thorac Surg. 2007 Nov;84(5):1508-13; discussion 1513-4. doi: 10.1016/j.athoracsur.2007.05.048. PMID 17954054
- [Background] O'Brien SM, Shahian DM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 2--isolated valve surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S23-42. doi: 10.1016/j.athoracsur.2009.05.056. PMID 19559823
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Rockville, MD. Calculating the U.S. Population-based EQ-5D Index Score: Research Initiative in Clinical Economics. February 2005. Agency for Healthcare Research and Quality, http://archive.ahrq.gov/professionals/clinicians-providers/resources/rice/EQ5Dscore.html
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Sousa-Uva M, Neumann FJ, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):4-90. doi: 10.1093/ejcts/ezy289. No abstract available. PMID 30165632
- [Background] Fujita B, Ensminger S, Bauer T, Mollmann H, Beckmann A, Bekeredjian R, Bleiziffer S, Schafer E, Hamm CW, Mohr FW, Katus HA, Harringer W, Walther T, Frerker C; GARY Executive Board. Trends in practice and outcomes from 2011 to 2015 for surgical aortic valve replacement: an update from the German Aortic Valve Registry on 42 776 patients. Eur J Cardiothorac Surg. 2018 Mar 1;53(3):552-559. doi: 10.1093/ejcts/ezx408. PMID 29190355